CLINICAL TRIAL: NCT03871374
Title: Factors Affecting Salt Intake in Young Adults
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: St Mary's University College (Other)
Responsible Party: Sponsor
Other Study IDs: SMEC_2018-19_007
Record Dates: First submitted 2019-03-04; First posted 2019-03-12 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Salt Intake

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
High salt intake is one of the key risk factors for development of high blood pressure and one of the main contributors to cardiovascular disease (CVD) mortality. Despite the efforts to reduce the intake of salt in the UK, current intake still exceeds the recommended values. It is evident that better understanding of this behaviour is necessary to be able to design more effective CVD prevention strategies. This study aims to explore the determinants of salt intake with the focus on genetics, salt taste perception and salt knowledge.

DETAILED DESCRIPTION:
Hypertension is a major cause of cardiovascular disease (CVD) and overall mortality. High dietary salt intake is a major risk factor for hypertension estimated to be responsible for one in ten deaths from CVD events. Salt consumption worldwide and in the UK exceeds the recommendations. One of the main determinants of food intake, and potentially salt, is taste which may be genetically determined. Research exploring the associations between genetics, salt taste and salt intake is scarce. Better understanding of these associations would be of specific interest in younger populations as it has been shown that it is the young adults that have higher preference for salty taste and consequently salt intake. Therefore, the aim of this study is to explore the associations between genetics, salt taste perception and salt intake in young UK adults.

One hundred participants (18-35 years) will be recruited. Salt taste thresholds will be identified using the British Standards Institution sensory analysis method (BS ISO 3972:2011) and preference for salty taste by rating the pleasantness and bitterness of six tomato soups with differing salt concentrations. Salt intake will be measured using five step multiple pass 24-hour recall completed via online platform (Online surveys) for one day of the week and one weekend day. Participants will be genotyped for genetic variants in the SCNN1B and TRPV1 genes coding for ion channels expressed in taste cells.

ELIGIBILITY:
Inclusion Criteria:

- Males or females, aged 18-35 years and healthy.

Exclusion Criteria:

* Current stage 1 or 2 hypertension
* Current or recent (less than one month prior to screening visit) use of antihypertensive medications or medications that affect BP
* Secondary hypertension
* History of cardiovascular disease, including myocardial infarction, congestive heart failure, stroke, and peripheral arterial disease
* Chronic kidney failure
* Peptic ulcer disease requiring treatment during the previous two years
* Currently pregnant women
* Underweight (BMI<18.5 kg/m2) and obese (BMI>30 kg/m2)
* Currently adhering to a low sodium diet
* Any illness that permanently alters taste
* Inability or unwillingness to participate or sign informed consent form
* Food allergy

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Hundred participants will be recruited based on their age and health status. In addition, this number is required to reach the adequate number of participants that has the genetic variation of interest (TRPV1 and SCNN1B genes).
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-03-15 (Estimated); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
Salt intake | 2 days observation
  Dietary salt intake - two 24-hour recalls

CONTACTS AND LOCATIONS:
Locations (1):
- St Mary's University, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No